CLINICAL TRIAL: NCT06854809
Title: Effects of Cognitive Functional Therapy Versus Therapeutic Exercises in Individuals With Chronic Shoulder Pain: A Randomized Controlled Trial
Brief Title: Cognitive Functional Therapy Versus Exercises for Chronic Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Matheus Dias Gregorio, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFTandShoulderPain
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Shoulder Pain
Keywords: shoulder pain; Psychosocial Rehabilitation; exercise therapy
MeSH Terms: conditions — Shoulder Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: This is a superiority randomized controlled trial, single-blinded, with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: Evaluators will be blinded to the treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive functional therapy (Experimental)
  Interventions: Behavioral: Cognitive functional therapy
- Therapeutic exercise (Active Comparator)
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Behavioral: Cognitive functional therapy — The intervention consists of a Cognitive-Functional Therapy (CFT) program for individuals with shoulder pain, conducted by trained physiotherapists (106 hours of training) under the supervision of an expert with over 8 years of experience. CFT adopts a biopsychosocial approach and is structured into three main components:
  Making Sense of Pain - A cognitive component aimed at reinterpreting dysfunctional beliefs about pain through a reflective process based on the patient's life history, promoting understanding and self-efficacy.
  Graded Exposure with Control - Gradual exposure to functional activities, aiming to modify maladaptive associations between movement and pain, fostering the development of movement confidence.
  Lifestyle Change - Discussion and implementation of strategies to promote a healthy lifestyle, including physical activity, sleep habits, and stress management.
  All three components are integrated from the first session, with initial focus on building the therapeutic all.
  Arms: Cognitive functional therapy
Other: Therapeutic exercise — Participants in the Therapeutic Exercises Group will engage in individualized exercises targeting the scapulothoracic musculature and rotator cuff. The exercises, performed bilaterally, include lateral arm rotation, T, W, wall hand slide, and diagonal arm movement upwards. Each participant will be guided by one of two physiotherapists, randomly assigned. The exercises will follow a protocol consisting of 3 sets of 12 repetitions, with 1-minute rest between sets, using progressively resistant Thera-Bands®. Resistance will increase when pain is ≤2 on the Numerical Rating Scale and perceived exertion is <3 on the Borg Scale. The protocol was designed based on scientific literature and shoulder pain treatment guidelines to address muscle activation deficits and rotator cuff and scapulothoracic imbalances.
  Arms: Therapeutic exercise

SUMMARY:
The objective of this clinical trial is to determine whether cognitive functional therapy is superior to therapeutic exercises for the treatment of chronic shoulder pain. The main questions it aims to answer are:

Is cognitive functional therapy superior to therapeutic exercises for pain and disability in individuals with chronic shoulder pain? Is cognitive functional therapy superior to therapeutic exercises for functionality and psychosocial factors?

Participants will:

Receive 4 to 8 sessions of cognitive functional therapy once a week for four to eight weeks.

Follow a therapeutic exercise protocol for eight weeks with a frequency of twice per week.

DETAILED DESCRIPTION:
This will be a randomized controlled trial, single-blind, with two parallel groups. 148 individuals with chronic shoulder pain will be randomly assigned to one of two groups: Cognitive functional therapy (CFT) or therapeutic exercises. The interventions will last between four and eight weeks, with the CFT group receiving therapy once a week and the therapeutic exercise group receiving sessions twice a week for eight weeks. The primary outcomes will be pain intensity and disability, while the secondary outcomes will include specific function, kinesiophobia, self-efficacy, sleep quality, treatment expectations, perception of change, treatment satisfaction and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

Individuals of both sexes, aged between 18 and 65 years, will be included if they have had shoulder pain for at least 3 months and report a pain intensity of at least 3 points on the Numeric Pain Rating Scale (NPRS) at rest or during arm movement. Additionally, they must have a minimum score of 20 points on the Shoulder Pain and Disability Index (SPADI).

Exclusion Criteria:

Individuals will not be included if they have adhesive capsulitis, defined as a loss of more than 50% of passive shoulder range of motion in external rotation; previous shoulder surgery; a history of shoulder fracture; systemic musculoskeletal diseases (e.g., rheumatoid arthritis, fibromyalgia); shoulder pain reproduced by active or passive cervical spine movement; signs of glenohumeral instability identified by a positive sulcus test or a positive apprehension test indicating laxity in the glenohumeral joint; self-reported systemic disease; a positive drop arm test; pregnancy; active cancer treatment; neurological diseases; cognitive impairments; corticosteroid injection within three months prior to the intervention; or physical therapy in the three months preceding the study.

Participants will be discontinued from the study if they experience fractures, surgeries, musculoskeletal or neural injuries that prevent access to treatment, or receive corticosteroid injections during the treatment or follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  The intensity of shoulder pain will be assessed during arm movement in which the patient reports, pain using the Numeric pain rating scale (NPRS). The scale consists of an 11-point ordinal system, ranging from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Shoulder disability | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Disability will be assessed using the Shoulder Pain and Disability Index (SPADI). The instrument is self-administered and consists of 13 items divided into 2 subscales (5 items for pain; 8 items for disability) and each item is scored from 0 to 10 points. The final score ranges from 0 to 100, with higher scores indicating greater shoulder disability.

SECONDARY OUTCOMES:
Patient Specific Function | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  The Patient Specific Functional Scale (PSFS) will be used to assess the patient's specific functionality. Patients will be asked to identify up to three important activities that they are having difficulty with or are unable to perform due to their condition. Furthermore, patients must classify, on a scale of 11 points (ranging from 0 "unable to perform activity" to 10 "able to perform activity".
Kinesiophobia | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Kinesiophobia will be assessed by the Tampa Kinesiophobia Scale 11 (TSK-11). The TSK is an instrument used to measure fear of movement. It is a self-administered questionnaire and presents 11 questions related to pain and intensity of symptoms. The score ranges from 11 to 44 points, in which higher scores indicate higher levels of kinesiophobia.
Pain Self-Efficacy | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Self-efficacy will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ). This is a 10-item self-report questionnaire that measures the degree of self-confidence in performing certain activities. Each item is rated on a 7-point Likert scale (0 = not at all confident; 6 = completely confident), with higher scores reflecting greater self-confidence.
Sleep Quality | Baseline, 4-week, at the end of treatment (8-week), and 12-week follow-up
  Sleep quality will be assessed using the Insomnia Severity Index (ISI). This is a scale that assesses the nature, intensity, and impact of insomnia experienced in the last month. The self-report instrument consists of 7 questions, answered using a Likert scale ranging from 0 (no severity) to 4 (high severity). The total score ranges from 0 to 28, classified as follows: no insomnia (0-7), mild insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28).
Expectations with Treatment | Baseline
  The patient's expectations regarding the treatment will be assessed by asking the question "How much do you expect your shoulder to improve at the end of the treatment?". The score will be measured on a 7-point Likert scale, with 1 being "worst possible" and 7 being "completely recovered". The assessment will be made before the intervention begins.
Perception of Change | 4-week, at the end of treatment (8-week), and 12-week follow-up
  The individual's perception of changes in health status over time will be measured using the Global Change Assessment Scale. The score varies from 15 points, with -7 being "a very significant worsening", 0 indicating "no change" and +7 "a very significant improvement"
Satisfaction with treatment | At the end of treatment (8-week), and 12-week follow-up
  The individual's satisfaction with the treatment will be measured using the Global Rating of Change Scale. The score varies from 15 points, with -7 being "the worst possible satisfaction", 0 indicating "no change" and +7 "the best possible satisfaction".
Exercise adherence | 4-week, at the end of treatment (8-week), and 12-week follow-up
  To assess exercise adherence, sections B and C of the Brazilian version of the Exercise Adherence Rating Scale (EARS-Br) will be used. Section B consists of 6 items rated on a 5-point Likert scale ranging from 0 ("strongly agree") to 4 ("strongly disagree"). This section aims to measure the participant's level of adherence to the recommended exercises. The total score ranges from 0 to 24 points, with scores equal to or greater than 17 indicating good adherence to the home exercise program. Section C consists of 9 items, also organized on a 5-point Likert scale (0 = "strongly agree"; 4 = "strongly disagree"). This section explores factors that influence exercise adherence, divided into barriers (items 1, 2, 3, 8, and 9) and facilitators (items 4, 5, 6, and 7).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sao Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared under request.
Supporting Information: Study Protocol, SAP
Time Frame: From December 1, 2027, to December 1, 2028, the data will be available for one year.
Access Criteria: The data will be shared with anyone who requests it via the responsible researcher's email.